CLINICAL TRIAL: NCT05438173
Title: A Randomized, Double-Blind, Crossover, Kinetic Study to Assess the Relative Bioavailability of Omega-3 Fatty Acids in Two Supplement Products in Healthy Adult Men and Women
Brief Title: Bioavailability of EPA/DHA in of Ruby-O and Krill Oil
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Center for Metabolic and Cardiovascular Research (Other)
Collaborators: Naturmega (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Other
Other Study IDs: MB-2201
Record Dates: First submitted 2022-06-24; First posted 2022-06-29 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: Bioavailability

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EPA + DHA Ruby-O (Experimental): Subject will receive a single 1000 mg oral dose of EPA + DHA Ruby-O capsule
  Interventions: Dietary Supplement: EPA + DHA Ruby-O
- EPA + DHA Krill Oil (Active Comparator): Subject will receive a single 1000 mg oral dose of EPA + DHA krill oil capsule
  Interventions: Dietary Supplement: EPA + DHA Krill Oil

INTERVENTIONS:
Dietary Supplement: EPA + DHA Ruby-O — Subject will receive a single 1000 mg oral dose of EPA + DHA Ruby-O capsule
  Arms: EPA + DHA Ruby-O
Dietary Supplement: EPA + DHA Krill Oil — Subject will receive a single 1000 mg oral dose of EPA + DHA krill oil capsule
  Arms: EPA + DHA Krill Oil

SUMMARY:
The objective of this study is to assess the relative bioavailability of eicosapentaenoic acid (EPA) and docosahexaenoic acid (DHA) in two supplement products in healthy adult men and women.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18 to 55 y of age, inclusive.
2. Subject has a BMI of 18.50 to 29.99 kg/m2.
3. Subject has a score ≥7 on the Vein Access Scale.
4. Subject is judged by the Investigator to be in generally good health, on the basis of medical history and screening measurements.
5. Subject is willing and able to undergo the scheduled study procedures.
6. Subject agrees to abstain from consuming more than one meal containing fish per week throughout the study.
7. Subject agrees to abstain from taking fish oil or omega-3 fatty acid supplements throughout the study.
8. Subject is willing to maintain usual physical activity levels for the duration of the study and not to engage in vigorous physical activity for at least 24 h prior to each clinic visit.
9. Subject is willing to abstain from alcohol consumption for at least 24 h prior to each clinic visit.
10. Subject has no plans to change smoking habits during the study.
11. Subject understands the study procedures and signs forms documenting informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has consumed more than one meal per week containing fish or seafood within 14 days prior to the first dose of study product (day 0) (washout is permitted).
2. Subject has taken a fish oil or omega-3 fatty acid supplement within 14 days prior to the first dose of study product (day 0) (washout is permitted).
3. Subject has consumed high-dose fish oil ≥1 g/d of EPA + DHA (the sum of EPA and DHA components from prescription or supplement forms) within 3 months prior to visit 2 (day 0).
4. Subject has consumed fish oil (prescription, dietary supplement, and/or EPA and/or DHA enriched foods) within 14 days of visit 2 (day 0).
5. Individual has used prescribed medication or over-the-counter medicinal products, including herbal and dietary supplements (EXCEPT for a daily omega-3 fatty acid-free vitamin and/or mineral supplement or the occasional use of acetaminophen or nonsteroidal anti-inflammatory drugs (such as ibuprofen or naproxen) within 14 days prior to visit 2 (day 0).
6. Subject has a laboratory test result of clinical significance based on the judgment of the Principal Investigator or qualified designee.
7. Subject has a positive result on the urine drug screen.
8. Subject has a clinically significant medical diagnosis that, in the opinion of the Investigator, could interfere with the interpretation of the study results.
9. Subject has uncontrolled hypertension (systolic blood pressure ≥160 mm Hg and/or diastolic blood pressure ≥100 mm Hg).
10. Subject has a recent history of cancer in the prior 2 years, except non-melanoma skin cancer or carcinoma in situ of the cervix.
11. Subject has signs or symptoms of an active infection of clinical relevance, or has taken antibiotics, within 14 days prior to any visit (washout is permitted).
12. Subject is a female who is pregnant, planning to be pregnant during the study period, lactating, or is of childbearing potential and is unwilling to commit to the use of a medically approved form of contraception throughout the study period.
13. Subject has a known allergy or sensitivity to any ingredients in the study products.
14. Subject has been exposed to any non-registered drug product within 30 days of the first screening visit.
15. Subject has a current or recent history (past 12 months of screening) or strong potential for illicit drug or excessive alcohol intake defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1.5 oz hard liquor).
16. Subject has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2022-07-11 (Actual); Primary Completion 2022-09-18 (Actual); Study Completion 2022-09-18 (Actual)

PRIMARY OUTCOMES:
Baseline-adjusted geometric mean ratio for EPA + DHA AUC | Baseline to 24 hours
  Changes in baseline-adjusted geometric mean ratio for EPA + DHA AUC

SECONDARY OUTCOMES:
Unadjusted maximum concentrations for EPA, DHA, and EPA + DHA | Baseline to 24 hours
  Changes in unadjusted maximum concentrations for EPA, DHA, and EPA + DHA
Unadjusted AUC for EPA, DHA, and EPA + DHA | Baseline to 24 hours
  Changes in unadjusted AUC for EPA, DHA, and EPA + DHA
Baseline-adjusted maximum concentration for EPA, DHA, and EPA + DHA | Baseline to 24 hours
  Changes in baseline-adjusted maximum concentration for EPA, DHA, and EPA + DHA
Baseline-adjusted AUC for EPA and DHA | Baseline to 24 hours
  Changes in baseline-adjusted AUC for EPA and DHA
Baseline-adjusted, dose-normalized maximum concentration for EPA, DHA, and EPA + DHA | Baseline to 24 hours
  Changes in baseline-adjusted, dose-normalized maximum concentration for EPA, DHA, and EPA + DHA
Baseline-adjusted, dose-normalized AUC for EPA, DHA, and EPA + DHA | Baseline to 24 hours
  Changes in baseline-adjusted, dose-normalized AUC for EPA, DHA, and EPA + DHA
Time to maximum concentration for EPA, DHA, and EPA + DHA | Baseline to 24 hours
  Changes in time to maximum concentration for EPA

CONTACTS AND LOCATIONS:
Overall Officials: Kevin C Maki, PhD, Study Director — MB Clinical Research & Consulting
Locations (1):
- Health Awareness, Port Saint Lucie, Florida, United States

IPD SHARING:
Plan to Share IPD: No